CLINICAL TRIAL: NCT06221605
Title: Probiotic Supplementation With BLa80, BL21, and LRa05 Stabilizes Lipid Metabolism in Chronic Hepatitis B Patients Receiving Tenofovir Alafenamide: A Clinical Trial
Brief Title: Composite Probiotics Stabilize Lipid Metabolism in Chronic Hepatitis B Patients:A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK2023009
Record Dates: First submitted 2024-01-11; First posted 2024-01-24 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): 30 billion CFU/sachet/day, before meals; Compound Probiotics (Bifidobacterium animalis subsp. animalis BLa80、Bifidobacterium longum subsp. longum BL21、Lacticaseibacillus rhamnosus LRa05) Storage: store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic
- placebo (Placebo Comparator): Maltodextrin, 1 sachet/day, before meals; Storage: store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — The intervention lasted for 3 months and 3 visits (at 0 month, 3rd and 6th month respectively).

SUMMARY:
The goal of this is to verify the clinical efficacy of compound probiotics in reducing HBV infection levels and regulating intestinal flora in patients with chronic hepatitis B.

The main question it aims to answer is:

• Conventional antiviral therapy combined with a 3-month probiotic intervention was used to evaluate the clinical efficacy of reducing HBV infection levels (HBeAg, HBsAg, and HBV DNA levels) and regulating gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the hepatitis B clinical diagnostic criteria of the Chronic Hepatitis B Prevention and Treatment Guidelines (2022 edition), excluding patients infected with hepatitis C virus, hepatitis D virus and other hepatitis viruses;
2. Be aware of the content and purpose of this study, and voluntarily sign the treatment study consent.

Exclusion Criteria:

1. Patients infected within 3 months;
2. Received antibiotic treatment within 3 months;
3. Received probiotic and probiotic therapy within 3 months;
4. Complicated with hypertension or diabetes;
5. Obesity or significantly low weight;
6. Obvious atherosclerosis;
7. Chronic kidney disease;
8. Inflammatory bowel disease, irritable bowel syndrome, or a history of gastrointestinal surgery;
9. Malignant tumors;
10. Autoimmune diseases;
11. Mental illnesses such as Parkinson's disease, Alzheimer's disease and stroke;
12. Pregnant or lactating women;
13. Patients with cirrhosis or decompensated liver disease;
14. Subjects cannot participate in the experiment due to their reasons; Those who meet any of the above criteria will not be selected.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Test the level of HBV infection in chronic hepatitis B patients | 6 months
  Evaluate HBsAg level in IU/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated with Fudan University, Shanghai, Shanghai Municipality, China